CLINICAL TRIAL: NCT01309867
Title: A Study to Evaluate the Performance of Two Designs of Soft Toric Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 680
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Toric Lens (Experimental): Bausch + Lomb investigational toric contact lenses
  Interventions: Device: Investigational Toric Lens
- PureVision Toric Lens (Active Comparator): Currently marketed Bausch + Lomb PureVision toric contact lenses
  Interventions: Device: PureVision Toric Lens

INTERVENTIONS:
Device: Investigational Toric Lens — Bausch & Lomb investigational toric contact lens worn on a daily wear basis for 2 weeks.
  Arms: Investigational Toric Lens
Device: PureVision Toric Lens — Currently marked Bausch & Lomb PureVision Toric Lens worn on a daily wear basis for 2 weeks.
  Arms: PureVision Toric Lens

SUMMARY:
The objective of the study is to evaluate the product performance of the Bausch + Lomb toric investigational contact lenses compared to the currently marketed PureVision toric contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have clear central corneas and be free of any anterior segment disorders.
* Subjects must be adapted lens wearers, wear a lens in each eye and each lens must be of the same manufacture and brand.
* Subjects must be myopic and require lens correction
* Subjects must be habitual wearers of toric soft contact lenses.

Exclusion Criteria:

* Subjects with any systemic disease currently affecting ocular health or which in the Investigator's opinion may have an effect on ocular health during the course of the study.
* Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Subjects with an active ocular disease or who are using any ocular medication.
* Subjects with any grade 2 or greater finding during the slit lamp examination. Subjects with corneal infiltrates, of ANY GRADE, are not eligible.
* Subjects with any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Subjects who are allergic to any component in the study care products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Barna, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 151 participants (302 eyes) were randomized to receive test contact lenses and 151 participants (302 eyes) were randomized to receive control contact lenses. After two weeks of wearing the first lens type, the participants crossed over to the second lens type for two weeks.
Groups:
- Investigational Toric Lens Then PureVision Toric Lens: Bausch + Lomb investigational toric contact lenses
  Investigational Toric Lens: Bausch & Lomb investigational toric contact lens worn on a daily wear basis for 2 weeks.
  Currently marketed Bausch + Lomb PureVision toric contact lenses PureVision Toric Lens: Currently marked Bausch & Lomb PureVision Toric Lens worn on a daily wear basis for 2 weeks.
- PureVision Toric Lens Then Investigational Toric Lens: Currently marketed Bausch + Lomb PureVision toric contact lenses
  PureVision Toric Lens: Currently marked Bausch & Lomb PureVision Toric Lens worn on a daily wear basis for 2 weeks.
  Bausch + Lomb investigational toric contact lenses Investigational Toric Lens: Bausch & Lomb investigational toric contact lens worn on a daily wear basis for 2 weeks.
Period: Overall Study
Arm/Group | Investigational Toric Lens Then PureVision Toric Lens | PureVision Toric Lens Then Investigational Toric Lens
Started | 151 | 151
Completed | 148 | 139
Not Completed | 3 | 12

BASELINE CHARACTERISTICS:
Population: A total of 151 participants were randomized to receive test contact lenses and 151 participants were randomized to receive control contact lenses. After two weeks of wearing the first lens type, the participants crossed over to the second lens type for two weeks.
Groups:
- All Participants: Participants were randomized 1:1 to receive test contact lenses or control contact lenses. After two weeks of wearing the first lens type, the participants crossed over to the second lens type for two weeks.
Arm/Group | All Participants
Number analyzed (Participants) | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 208
  Male | 94

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Absolute Lens Rotation ≤ 10 Degrees.
Time Frame: 2 weeks
Population: There were 518 eyes in each group for this outcome measure.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Toric Lens | PureVision Toric Lens
Number analyzed (Participants) | 259 | 259
Number analyzed (eyes) | 518 | 518
eyes | 489 | 426

2. Primary Outcome: Visual Acuity
Description: Visual acuity was assessed by distance high contrast logarithm of the minimum angle of resolution (logMAR).
Time Frame: 2 weeks
Population: There were 518 eyes in each group for this outcome measure.
Measure: Least Squares Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Investigational Toric Lens | PureVision Toric Lens
Number analyzed (Participants) | 259 | 259
Number analyzed (eyes) | 518 | 518
logMAR | -0.025 (0.106) | -0.021 (0.106)

3. Secondary Outcome: Symptoms and Complaints
Description: Symptoms/complaints were assessed on a scale from 0 to 100, with 0 denoting unfavorable symptoms/complaints. Symptoms/complaints were recorded at each post-dispensing visit based on the subject's experience with the study lens worn prior to the visit. The symptoms/complaints parameters were: Burning/stinging upon insertion; Comfort upon insertion, Overall comfort, and Comfort at the end of the day; Ease of handling/insertion, and Ease of handling/removal; Dryness; Itchiness; Redness; Vision; Lens cleanliness; and Overall impression.
Time Frame: 2 weeks
Population: There were 571 eyes in each group assess for this outcome measure.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Investigational Toric Lens | PureVision Toric Lens
Number analyzed (Participants) | 286 | 286
Number analyzed (eyes) | 571 | 571
score on a scale
  Burning/stinging upon insertion | 85.4 (28.1) | 82.0 (28.1)
  Comfort upon insertion | 77.7 (29.4) | 74.3 (29.4)
  Overall comfort | 77.3 (29.6) | 67.9 (29.6)
  Comfort at the end of the day | 67.8 (33.6) | 57.6 (33.6)
  Ease of handling/insertion | 84.4 (25.2) | 80.9 (25.2)
  Ease of handling/removal | 87.6 (23.0) | 83.7 (23.0)
  Dryness | 73.6 (32.1) | 66.3 (32.1)
  Itchiness | 86.6 (26.0) | 82.0 (26.0)
  Redness | 88.0 (23.9) | 83.5 (23.9)
  Vision | 82.0 (28.3) | 73.9 (28.3)
  Lens Cleanliness | 86.1 (22.1) | 83.5 (22.1)
  Overall impression | 74.4 (30.3) | 64.2 (30.3)

4. Secondary Outcome: Percentage of Eyes With > Grade 2 Slit Lamp Findings
Description: Graded slit lamp findings for each eye, including epithelial edema, epithelial microcysts, corneal staining, limbal and bulbar injections, upper lid tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates were graded for severity on a scale from 0 (No Finding) to 4 (Severe Finding). The outcome measure is any finding > grade 2, across abnormalities.
Time Frame: 2 weeks
Population: There were 600 eyes with non-missing scores in both groups for this outcome measure.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Toric Lens | PureVision Toric Lens
Number analyzed (Participants) | 300 | 300
Number analyzed (eyes) | 600 | 600
eyes | 1 | 1

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Adverse events were not coded. Therefore, source vocabulary is not applicable. There were 302 eyes dispensed each lens group, assessed for adverse events.
Arm/Group | Investigational Toric Lens | PureVision Toric Lens
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/151
Other Adverse Events (participants affected / at risk) | 0/151 | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.